CLINICAL TRIAL: NCT05605145
Title: Pneumocystis Pneumonia in Immunocompromised Population in Southern China：A Multicenter,Open,Prospective Study
Brief Title: PCP in Immunocompromised Population in Southern China
Acronym: PCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: People's Hospital of Guangxi Zhuang Autonomous Region (Other); The Fourth People's Hospital of Nanning (Other); Chest Hospital of Guangxi Zhuang Autonomous Region (Unknown); People's Hospital of Baise (Unknown); LiuZhou People's Hospital (Other); The second Nanning People's Hospital (Unknown); The People's Hospital of Wuzhou (Unknown); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); 923rd Hospital of the People's Liberation Army (Unknown)
Responsible Party: Sponsor
Other Study IDs: GX-PCP-2020
Record Dates: First submitted 2022-10-10; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Immunocompromised Patients; Pneumocystis Pneumonia; Diagnosis; Polymerase Chain Reaction
Keywords: Pneumocystis Pneumonia; Immunocompromised Patients; Polymerase Chain Reaction; Treatment
MeSH Terms: conditions — Pneumonia, Pneumocystis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Respiratory tract specimens such as alveolar lavage fluid, sputum and throat swabs were collected from all patients who met the enrollment conditions of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunocompromised patients: 1. Patients with immunocompromised conditions, including but not limited to HIV infection, long-term systemic use of corticosteroids, use of immunosuppressive agents, hematologic malignancies, solid tumors, hematopoietic stem cell transplantation, solid organ transplantation, radiotherapy and/or chemotherapy for malignancies,primary immunodeficiency disease.
  2. Typical clinical manifestations of PJP such as fever,nonproductive cough, shortness of breath, and progressive hypoxemia.
  3. Radiological abnormalities suggestive to PJP in bilateral lungs revealed by chest computed tomography (CT).
  4. Respiratory tract samples were collected for qPCR and/or mNGS detection.
  Interventions: Diagnostic Test: PCR was used to detect pneumocystis in respiratory specimens

INTERVENTIONS:
Diagnostic Test: PCR was used to detect pneumocystis in respiratory specimens — Respiratory tract specimens such as alveolar lavage fluid, sputum and throat swabs were collected from all patients who met the enrollment conditions of this study. qPCR and/or mNGS were used to detect pneumocystis in respiratory specimens.

SUMMARY:
To evaluate the sensitivity and specificity of the combined detection system for the diagnosis of pneumocystis infection in immunocompromised population in Southern China.

DETAILED DESCRIPTION:
Pneumocystis jirovecii pneumonia (PJP) is a serious opportunistic infection in immunocompromised patients, with a difficult diagnosis, rapid progression and high mortality rate. The PJP mortality rate is high among patients with delayed diagnosis and treatment, and death is due to severe respiratory failure. Up to now, data regarding Pneumocystis jirovecii infection in immunocompromised patients is limited. In the present prospective study, the investigators aimed to evaluate the sensitivity and specificity of the combined detection system for the diagnosis of pneumocystis infection in immunocompromised population in Southern China.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with immunocompromised conditions, including but not limited to HIV infection, long-term systemic use of corticosteroids, use of immunosuppressive agents, hematologic malignancies, solid tumors, hematopoietic stem cell transplantation, solid organ transplantation, radiotherapy and/or chemotherapy for malignancies,primary immunodeficiency disease.
2. Patients with typical clinical manifestations of PJP such as fever,nonproductive cough, shortness of breath, and progressive hypoxemia.
3. Patients with radiological abnormalities suggestive to PJP in bilateral lungs revealed by chest computed tomography (CT).
4. Respiratory tract samples were collected for qPCR and/or mNGS detection.

Exclusion Criteria:

1. Patients who were unable to obtain a respiratory specimen.
2. Medical record was incomplete.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Immunocompromised patients who have fever, respiratory symptoms or pulmonary imaging changes were recruited into group.Respiratory tract specimens such as alveolar lavage fluid, sputum and throat swabs were collected from enrolled patients and detected for pneumocystis by the combined detection system including qPCR and/or mNGS.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
PJP diagnosis rate | 1 week
  Proven pneumocystis jirovecii pneumonia（PJP）was defined as direct microscopy positive finding of a bronchopulmonary specimen. The diagnosis of probable PJP was applied to patients with a positive qPCR or metagenomic Next-Generation Sequencing（mNGS）and several criteria including an underlying immunosuppressive condition, clinical symptoms and radiological signs deemed to be compatible with PJP by clinicians. Pneumocystis jirovecii colonization was defined as any case presented with a positive qPCR or mNGS, which was not included in the previous two groups. Non-PjP corresponded to a negative Pj result by the above detection method(direct microscopy,qPCR or mNGS).

SECONDARY OUTCOMES:
Treatment response rate of PJP | 3 months
  Treatment response was defined as one of the followings: (1)amelioration or resolution of baseline signs and symptoms, chest computed tomography (CT), and hospital discharge; (2)clinical improvement sustained at least 2 to 4 weeks after cessation of antifungal therapy.
Overall Survival rate | 3 months
  Survival was defined as being alive 3 months after symptoms onset.

CONTACTS AND LOCATIONS:
Overall Officials: Cunwei Cao, MD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No